CLINICAL TRIAL: NCT02592356
Title: Effects of Tyrosine Kinase Inhibitors on Body Composition in Endocrine Tumors -- A Pilot Study
Brief Title: Effect of Cabozantinib S-Malate or Lenvatinib Mesylate on Weight and Body Composition in Patients With Metastatic Endocrine Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0864; NCI-2015-02058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0864 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-10-27; First posted 2015-10-30 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Differentiated Thyroid Gland Carcinoma; Malignant Adrenal Gland Pheochromocytoma; Malignant Paraganglioma; Thyroid Gland Medullary Carcinoma
MeSH Terms: conditions — Paraganglioma, Extra-Adrenal; Carcinoma, Medullary | interventions — Absorptiometry, Photon; Restraint, Physical; cabozantinib; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib or Lenvatinib (Experimental): Patients treated with cabozantinib s-malate or lenvatinib mesylate are observed for body weight, skeletal muscle and adipose tissue changes. Patients complete 3 to 4 questionnaires every 2 weeks for 6 months and then monthly up to 12 months. Patients also undergo physical assessments and body composition measurements by DXA and CT scans at baseline, months 3, 6, and 12.
  Interventions: Procedure: Computed Tomography; Procedure: Dual X-ray Absorptiometry; Procedure: Physical Examination; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Cabozantinib; Drug: Lenvatinib

INTERVENTIONS:
Procedure: Computed Tomography — Correlative studies
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Dual X-ray Absorptiometry — Correlative studies
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Procedure: Physical Examination — Correlative studies
  Other Names: assessment; Physical; Physical Assessment; PHYSICAL EXAM
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Cabozantinib
  Other Names: XL-184; XL184
Drug: Lenvatinib
  Other Names: E7080; Lenvima

SUMMARY:
The goal of this clinical research study is to learn about possible weight, muscle, and/or fat loss in patients receiving cabozantinib or lenvatinib.

DETAILED DESCRIPTION:
Baseline Visit

If you agree to take part in this study, you will have the following tests and procedures at a baseline visit within 10 days after starting either cabozantinib or lenvatinib:

Your height, weight, waist, and hips will be measured. You will have basic tests of your physical strength and balance. Your hand grip strength will be measured, you will be asked to rise from a chair without using your arms to push off, and you will complete a 6-minute walk test.

You will have a full-body dual-energy x-ray absorptiometry (DXA) scan to measure the amount of fat and muscle in your body. Images from a standard computed tomography (CT) scan will also be collected and reviewed for this purpose. If you are scheduled only for a chest CT scan as part of your regular care, your abdomen will also be scanned at the same time for research purposes.

You will meet with a dietician to talk about your current and past eating habits.

You will fill out questionnaires about any pain or other symptoms you may have had; about any gastrointestinal (GI) side effects you may be having before you start chemotherapy; about the amount of physical exercise and activity you get; and about your food intake over the last 24 hours. Together the questionnaires should take about 20-25 minutes to complete.

You will be receiving cabozantinib or lenvatinib as part of your standard of care.

Study Visits After the baseline visit, you will have study visits on the following schedule. Some of these visits will be at the same time as your scheduled clinic visits with your regular doctor. However, some assessments will be done in between clinic visits online or by phone.

Month 1 and 2:

One (1) time every 2 weeks (+/- 1 week) during Months 1 and 2, you will fill out 3 questionnaires at home:

You will be asked about any gastrointestinal (GI) and other side effects you may be having. This will be done by phone and should take about 5-10 minutes.

You will fill out an online questionnaire at home about your eating habits over the last 24 hours. If you do not have internet access, you will complete the questionnaire over the phone with a member of the study staff. This should take about 10 minutes.

You will complete a questionnaire about any symptoms you may be having online or by phone. This should take about 5-8 minutes.

At Months 3, 6, and 12 (± 4 weeks) you will come to the clinic:

Your height, weight, waist, and hips will be measured. You will have the same tests of your physical strength and balance that you had at the baseline visit.

You will complete the same questionnaires you completed at the baseline visit. These will be done on paper or on a computer or tablet.

You will have a DXA scan to measure the amount of fat and muscle in your body. If you are having certain GI side effects (such as diarrhea, nausea, vomiting, mouth sores, and so on), the study doctor will talk with you about receiving standard drugs to help with those side effects. You may ask the study staff for information about how the drugs are given and their risks. You may also meet with a dietician, who may recommend ways to help improve some side effects.

Between clinic visits:

Two (2) times per month (+/- 1 week) between Months 3 and 6, and once a month (+/- 1 week) between Months 6 and 12, you will complete 3 questionnaires at home about your food intake over the past 24 hours; any symptoms you may be having; and any GI or other side effects you may be having. The questionnaires may be completed online or by phone and together should take about 20 minutes.

Length of Study Participation Your participation in this study will be over after the Month 12 visit

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Initiating cabozantinib for progressive DTC, MTC, malignant PH or PGs or lenvatinib for progressive DTC or MTC as determined by patient's endocrinologist
* ECOG performance status 0-2
* Able to communicate in English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* Active participation in any weight reduction program including use of drugs used for weight loss
* Inability to ambulate without assistance (e.g. cane, walker)
* Multiple Endocrine Neoplasia (MEN) 2B (due to differences in body habitus)
* Patients unwilling or unable to comply with the protocol.
* Use of chronic (>3 months consecutively) non-physiological (15 mg/m² hydrocortisone equivalent) doses of glucocorticoids
* Non-English speaking PH and PG patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in weight among patients who have no gastrointestinal (GI) adverse events (AEs) or have =< grade 1 symptoms and those with grade 2 or above AEs, according to the National Cancer Institute Common Toxicity Criteria version 4.0 | Baseline to up to 6 months
  2-sided paired t-test will be used to measure weight change after successful intervention of diarrhea and anorexia. Linear mixed-effects model will be used to explore the longitudinal weight changes. Summary descriptive statistics, including proportions, medians, means, 95% confidence intervals, and other simple statistics will be provided for demographics, gastrointestinal adverse events, body composition changes and blood markers. 95% confidence intervals (CI) will be reported for the accuracy of DXA compared to computed tomography CT. The correlation between change of weight/body composition and tumor response will be investigated by logistic regression.

SECONDARY OUTCOMES:
Change in weight in patients with metastatic endocrine tumors during active intervention to control diarrhea and anorexia | Baseline to up to 12 months
  Summary descriptive statistics, including proportions, medians, means, 95% confidence intervals, and other simple statistics will be provided for demographics, body composition changes and blood markers. 95% CI will be reported for the accuracy of DXA compared to CT. The correlation between change of weight/body composition and tumor response will be investigated by logistic regression.
Change in adipose tissue in patients with metastatic endocrine tumors during active intervention to control diarrhea and anorexia | Baseline to up to 12 months
  Summary descriptive statistics, including proportions, medians, means, 95% confidence intervals, and other simple statistics will be provided for demographics, body composition changes and blood markers. 95% CI will be reported for the accuracy of DXA compared to CT. The correlation between change of weight/body composition and tumor response will be investigated by logistic regression.
Change in skeletal muscle in patients with metastatic endocrine tumors during active intervention to control diarrhea and anorexia | Baseline to up to 12 months
  Summary descriptive statistics, including proportions, medians, means, 95% confidence intervals, and other simple statistics will be provided for demographics, body composition changes and blood markers. 95% CI will be reported for the accuracy of DXA compared to CT. The correlation between change of weight/body composition and tumor response will be investigated by logistic regression.

OTHER OUTCOMES:
Tumor response | Up to 12 months
  Summary descriptive statistics, including proportions, medians, means, 95% confidence intervals, and other simple statistics will be provided for demographics, tumor response rates and blood markers. 95% CI will be reported for the accuracy of DXA compared to CT. The correlation between change of weight/body composition and tumor response will be investigated by logistic regression.
Quality of life change | Baseline to up to 12 months
  Summary descriptive statistics, including proportions, medians, means, 95% confidence intervals, and other simple statistics will be provided for demographics, tumor response rates and blood markers. 95% CI will be reported for the accuracy of DXA compared to CT. The correlation between change of weight/body composition and tumor response will be investigated by logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Naifa L Busaidy, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org